CLINICAL TRIAL: NCT06826014
Title: Texas Regional Excellence in Cancer (TREC) @Texas A&M University Cancer Prevention Registry and Repository
Brief Title: TREC@TAMU Cancer Prevention Registry and Repository
Status: Recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY2024-0008
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Genetics; Disease; Diet; Lifestyle Factors
Keywords: cancer; genetics
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood, urine, saliva, and/or cheek cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study collects health and genetic information to implement cancer prevention and treatment strategies.

DETAILED DESCRIPTION:
This research will explore how genetics, diet, exercise, and jobs influence the risk of developing cancers that can be treated early. The goal is to find out if this knowledge can help doctors and health insurers improve their methods for preventing cancers that cannot be treated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, and,
* People participating in the Cancer Prevention and Research Institute of Texas (CPRIT) A coordinated cancer screening research program in Bryan and Navasota Family Medicine Clinics and,
* People with COPD, liver disease, cervical intraepithelial neoplasia (CIN) lesions, having had a colonoscopy or a low dose computed tomography (LDCT) lung scan or cervical exam in the last 12 months or scheduled for one, and,
* Able to give and comprehend the consent process, and,
* Able to consent to donate blood and urine samples, genetic material through buccal swabs for future research, and,
* Able to understand that their specimens, health record, and changes in health status will be followed for a five-year period and shared in deidentified form with the research community, and,
* All sexes and gender identities.

Exclusion Criteria:

* Declines to participate or interact with staff/share their medical status.
* A diagnosis of Alzheimer's disease or related dementias in a medical record indicates a progressive, debilitating condition that impairs memory, thought processes, and functioning Individuals who are unable or unwilling to provide consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TREC@TAMU Registry will recruit as many participants as possible. The estimated enrollment in five years is expected to be 2500, but investigators will not limit recruitment if that number is exceeded.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and nature of ADRs on the Naranjo Scale Questionnaire | 5 years
  Measure the frequency and nature of adverse drug reactions by obtaining a complete medical history and physical examination and validating the patient's current concomitant medication list during the office visit. Patient medical information would be input into the ActX platform, which functions as a computable EHR medical record analysis, evaluation of polypharmacy status, and monitoring of ADRs using the Naranjo Scale will be conducted for the duration of the study.

SECONDARY OUTCOMES:
Self-reported Health status and any significant changes | 5 years
  The EQ-5D-5L survey, designed to collect data on health status and significant changes, will be administered to every patient in the registry at each clinic visit and at least every six months for five years after enrollment.
  The EQ-5D-5L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension features five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Patients indicate their health state by ticking the box next to the most appropriate statement for each dimension. This choice generates a one-digit number representing the selected level for that dimension. The numbers from the five dimensions can be combined into a five-digit number that characterizes the patient's health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M Family Care, Bryan, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT06826014/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT06826014/SAP_001.pdf